CLINICAL TRIAL: NCT01669772
Title: Study on the Effects of DA-9701 on Gastrointestinal Motility on Healthy Adult Males and Female Subjects
Brief Title: Study on the Effects of DA-9701 on Gastrointestinal Motility on Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Myung-gui Choi (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Myung-gui Choi, Professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA-9701 trial
Record Dates: First submitted 2012-08-12; First posted 2012-08-21 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — DA-9701

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DA-9701 and placebo (Other): Administer DA-9701 for 1week and assess the study outcomes. After 1 week of washout period, administer placebo for 1week and assess the outcomes again.
  Interventions: Drug: DA-9701 and placebo
- Placebo and DA-9701 (Other): Administer placebo for 1 week and study the outcome parameters. After 1 week of washout, administer DA-9701 for 1 week and assess the outcome parameters again.
  Interventions: Drug: Placebo and DA-9701

INTERVENTIONS:
Drug: DA-9701 and placebo — Prescribe 30mg of DA-9701(motilitone) t.i.d for 1 week and then crossover to placebo.
  Other Names: DA-9701(motilitone)
  Arms: DA-9701 and placebo
Drug: Placebo and DA-9701 — Administer placebo 1 tablet t.i.d for 1 week. After 1 week of washout, crossover to 30mg of DA-9701 t.i.d. for 1 week.
  Other Names: DA-9701(motilitone)
  Arms: Placebo and DA-9701

SUMMARY:
DA-9701 is a new prokinetic agent formulated with Pharbitis Seed and Corydalis Tuber. These plants have been used in oriental traditional medicine for the treatment of gastrointestinal maladies. In a stage 3 trial, its' efficacy has been compared to that of itopride in functional dyspepsia patients and proved to have comparable safety and efficacy. However, its' exact effect on the gastrointestinal motility has not been completely elucidated. This study will study the effects of DA-9701 on the healthy adult gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults of either sex, at least 20 years of age
* Having no abdominal discomfort or pain
* No diseases diagnosed by screening gastroduodenoscopy
* Having given voluntary written consent

Exclusion Criteria:

* Currently participating or having participated in another drug trial within four weeks of trial start.
* Women of childbearing age who are either pregnant, breast-feeding or not under proper contraceptive methods.
* A history of surgery which may affect gastrointestinal motility.
* Subjects with gastrointestinal bleeding, mechanical obstruction or perforation.
* Subjects with irritable bowel syndrome or inflammatory bowel disease.
* Subjects with serious conditions involving the liver, kidneys, heart, lung or endocrinology system.
* Psychiatric disease patients, substance abuse subjects such as alcohol or drugs.
* Subjects who have taken drugs that may affect the study outcome such as antibiotics, corticosteroids or NSAIDS within 1 month or motility agents, H2 receptor blockers, proton pump inhibitors, anticholinergics, erythromycin or antipsychotics within 2 weeks.
* Other reasons that the investigator considers valid.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Study the effects of DA-9701 on GI motility in healthy adult volunteers | 3weeks
  Study the effects of DA-9701 on gastrointestinal motility in healthy adult volunteers

SECONDARY OUTCOMES:
Examine the effects of DA-9701 by Scintigraphic transit measurement | 3weeks
  Examine the effects of DA-9701 by Scintigraphic transit measurement
Examine the effects of DA-9701 by EGG/Drink test | 3weeks
  Examine the effects of DA-9701 by EGG/Drink test
Examine the effects of DA-9701 by SPECT | 3weeks
  Examine the effects of DA-9701 by SPECT

CONTACTS AND LOCATIONS:
Overall Officials: Myong Ki Baeg, MD, Principal Investigator — CU Korea, Seoul St Mary's Hospital
Locations (1):
- Seoul St Mary's hospital, Seoul, South Korea